CLINICAL TRIAL: NCT01495611
Title: Predicting Perioperative Opioid Adverse Effects and Personalizing Analgesia in Children: A Multicenter Pharmacogenetic Study
Brief Title: Multicenter Perioperative Opioid Pharmacogenetic Study
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Baylor College of Medicine (Other); Ochsner Health System (Other); Children's Hospital Colorado (Other); Children's Hospital Los Angeles (Other); C.S. Mott Children's Hospital (Other); St. Christopher's Hospital for Children (Other); St. Louis Children's Hospital (Other); Boston Children's Hospital (Other); Seattle Children's Hospital (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Wisconsin, Madison (Other); University of Miami (Other); Johns Hopkins University (Other); Stanford University (Other); Phoenix Children's Hospital (Other); University of Michigan (Other); University of Utah (Other); Shanghai Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-1353
Record Dates: First submitted 2011-12-12; First posted 2011-12-20 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pain
Keywords: postoperative,; pediatric; pharmacogenetic; opioid; morphine; perioperative; respiratory depression
MeSH Terms: conditions — Pain; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A database/ repository will be constructed for future research, analysis, and recruitment. De-identified study subjects' genetic information and their responses to pain and pain medications, side-effects will be included in the database. Blood specimens will be included in the repository for exploring potentially important SNPs and biomarkers in future. No patient identifiers will be included in the repository and there will be a confidential (access limited to investigators only) code or link between the repository/database and other information about the participant.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to identify factors and genes (the DNA material that determines the makeup of the human body) that may be associated with how children respond to pain medication. Specifically, the investigators want to study factors that may be associated with pain sensitivity, morphine requirement after surgery and side-effects from morphine and other pain medications. The investigators expect that the information obtained in this research study will help us to develop more effective, safe, and tailored treatment options in the future.

DETAILED DESCRIPTION:
Opioid drugs as a group have withstood the test of time in their ability to relieve pain. Morphine is the most frequently used "gold standard" opioid for managing surgical pain. Like other opioids, morphine has a narrow therapeutic index and a large inter-patient variability in response. Certain genetic and non-genetic factors are believed to be responsible for variations in analgesic responses and side effects with morphine. Genetic factors determining an individual's pain sensitivity and regulating morphine's pharmacokinetics (transporters) and pharmacodynamics (receptors and signal transduction elements) are likely contributors to such variability. Frequent variations in analgesic response are unfortunately clinically significant with inadequate pain relief at one end of the spectrum of responses and major side effects including potentially fatal respiratory depression due to relative overdosing at the other end. Much of the inter-individual variability in response to a dose of morphine following surgical procedures can be explained by single nucleotide polymorphisms (SNPs) in a subset of the genes that encode proteins involved in pain perception, opioid transport and opioid receptor signaling. The genetic variants of mu opioid receptor (OPRM1), Catechol-O-methyltransferase (COMT), the Multi Drug Resistance Transport protein gene ABC B1, have been associated in small adult studies with varying levels of pain sensitivity, analgesic response to opioids and susceptibility to serious side-effects of opioids such as respiratory depression, sedation and vomiting. Effective and safe acute postoperative pain relief in a subset of children is clinically difficult due to frequent clinical variations in perceptions of pain and responses to opioids. To the investigator's knowledge, there is no other study attempting to individualize perioperative analgesia in children. The investigator's long term goal is to identify factors that modify pain sensitivity and responses to morphine in order to develop more effective, safe and tailored therapies. The overall objective of this application is to evaluate the contribution of individual and combined affects of genetic polymorphisms in OPRM1, COMT and ABC B1 genes and their association with postoperative pain relief and adverse effects with morphine. The investigator's central hypothesis is that specific genetic polymorphisms in genes involved in pain perception, opioid transport and opioid receptor signaling pathways contribute significantly to pain sensitivity, morphine consumption, and morphine's side-effects in children.

This study will also explore a set of other important SNPs that might influence pain perception and responses to morphine in children. The data will be analyzed looking at pain scores, morphine doses, incidence of side-effects of morphine including respiratory depression, sedation, vomiting and itching.

ELIGIBILITY:
Inclusion Criteria:

* children 6-17 years of age
* ASA physical status 1 and 2
* scheduled for tonsillectomy (T) and tonsillectomy and adenoidectomy (T and A)
* Children with obstructive sleep apnea will also be included.

Exclusion Criteria:

* children with developmental delay
* liver and renal diseases,
* preoperative pain requiring analgesics (e.g. chronic tonsillitis).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing adenotonsillectomy in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2017-04-30

PRIMARY OUTCOMES:
Safety Outcomes | Post-anesthetic recovery room, an expected average of 2 hours
  Incidence of serious opioid related adverse effects including respiratory depression, excessive sedation, nausea and vomiting in recovery room.

SECONDARY OUTCOMES:
Efficacy Outcome Measures - Opioid interventions | Post-anesthetic recovery room, an expected average of 2 hours
  Number of opioid interventions required in the recovery room
Efficacy Outcome Measures - Opioid requirement | Post-anesthetic recovery room, an expected average of 2 hours
  Total opioid requirement will be measured
Efficacy Outcome Measures - Pain Scores | Post-anesthetic recovery room, an expected average of 2 hours
  Pain scores as measured by the Numerical Rating Scale (NRS) and the Facial expression, Leg movement, Activity, Cry, and Consolability (FLACC) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Sadhasivam, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (15):
- United States (15):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - The Children's Hospital, Denver, Denver, Colorado
  - University of Miami - Miller School of Medicine, Miami, Florida
  - Children's Memorial Hospital, Chicago, Illinois
  - Ochsner Medical Center for Children, New Orleans, Louisiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - UW Health-American Family Children's Hospital, Madison, Wisconsin

REFERENCES:
- [Background] Diatchenko L, Slade GD, Nackley AG, Bhalang K, Sigurdsson A, Belfer I, Goldman D, Xu K, Shabalina SA, Shagin D, Max MB, Makarov SS, Maixner W. Genetic basis for individual variations in pain perception and the development of a chronic pain condition. Hum Mol Genet. 2005 Jan 1;14(1):135-43. doi: 10.1093/hmg/ddi013. Epub 2004 Nov 10. PMID 15537663
- [Background] Chou WY, Wang CH, Liu PH, Liu CC, Tseng CC, Jawan B. Human opioid receptor A118G polymorphism affects intravenous patient-controlled analgesia morphine consumption after total abdominal hysterectomy. Anesthesiology. 2006 Aug;105(2):334-7. doi: 10.1097/00000542-200608000-00016. PMID 16871067
- [Background] Oertel BG, Schmidt R, Schneider A, Geisslinger G, Lotsch J. The mu-opioid receptor gene polymorphism 118A>G depletes alfentanil-induced analgesia and protects against respiratory depression in homozygous carriers. Pharmacogenet Genomics. 2006 Sep;16(9):625-36. doi: 10.1097/01.fpc.0000220566.90466.a2. PMID 16906017
- [Background] Sutters KA, Miaskowski C. Inadequate pain management and associated morbidity in children at home after tonsillectomy. J Pediatr Nurs. 1997 Jun;12(3):178-85. doi: 10.1016/S0882-5963(97)80075-9. PMID 9198341
- [Background] Sutters KA, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Savedra MC, Lanier B. A randomized clinical trial of the effectiveness of a scheduled oral analgesic dosing regimen for the management of postoperative pain in children following tonsillectomy. Pain. 2004 Jul;110(1-2):49-55. doi: 10.1016/j.pain.2004.03.008. PMID 15275751
- [Background] Hamers JP, Abu-Saad HH. Children's pain at home following (adeno) tonsillectomy. Eur J Pain. 2002;6(3):213-9. doi: 10.1053/eujp.2001.0326. PMID 12036308
- [Background] Homer JJ, Frewer JD, Swallow J, Semple P. An audit of post-operative analgesia in children following tonsillectomy. J Laryngol Otol. 2002 May;116(5):367-70. doi: 10.1258/0022215021910807. PMID 12080995
- [Background] Homer JJ, Swallow J, Semple P. Audit of pain management at home following tonsillectomy in children. J Laryngol Otol. 2001 Mar;115(3):205-8. doi: 10.1258/0022215011907208. PMID 11244527
- [Background] Huth MM, Broome ME. A snapshot of children's postoperative tonsillectomy outcomes at home. J Spec Pediatr Nurs. 2007 Jul;12(3):186-95. doi: 10.1111/j.1744-6155.2007.00111.x. PMID 17594298
- [Background] Huth MM, Broome ME, Good M. Imagery reduces children's post-operative pain. Pain. 2004 Jul;110(1-2):439-48. doi: 10.1016/j.pain.2004.04.028. PMID 15275797
- [Background] Gedaly-Duff V, Ziebarth D. Mothers' management of adenoid-tonsillectomy pain in 4- to 8-year-olds: a preliminary study. Pain. 1994 Jun;57(3):293-299. doi: 10.1016/0304-3959(94)90004-3. PMID 7524009
- [Background] Warnock FF, Lander J. Pain progression, intensity and outcomes following tonsillectomy. Pain. 1998 Mar;75(1):37-45. doi: 10.1016/S0304-3959(97)00202-9. PMID 9539672
- [Background] Burkart CM, Steward DL. Antibiotics for reduction of posttonsillectomy morbidity: a meta-analysis. Laryngoscope. 2005 Jun;115(6):997-1002. doi: 10.1097/01.MLG.0000163749.77019.8F. PMID 15933509
- [Background] Perquin CW, Hazebroek-Kampschreur AAJM, Hunfeld JAM, Bohnen AM, van Suijlekom-Smit LWA, Passchier J, van der Wouden JC. Pain in children and adolescents: a common experience. Pain. 2000 Jul;87(1):51-58. doi: 10.1016/S0304-3959(00)00269-4. PMID 10863045
- [Background] Duedahl TH, Hansen EH. A qualitative systematic review of morphine treatment in children with postoperative pain. Paediatr Anaesth. 2007 Aug;17(8):756-74. doi: 10.1111/j.1460-9592.2007.02213.x. PMID 17596221
- [Background] Anderson BJ, Palmer GM. Recent developments in the pharmacological management of pain in children. Curr Opin Anaesthesiol. 2006 Jun;19(3):285-92. doi: 10.1097/01.aco.0000192802.33291.6f. PMID 16735812
- [Background] Klepstad P, Dale O, Skorpen F, Borchgrevink PC, Kaasa S. Genetic variability and clinical efficacy of morphine. Acta Anaesthesiol Scand. 2005 Aug;49(7):902-8. doi: 10.1111/j.1399-6576.2005.00772.x. PMID 16045647
- [Background] Berde CB, Sethna NF. Analgesics for the treatment of pain in children. N Engl J Med. 2002 Oct 3;347(14):1094-103. doi: 10.1056/NEJMra012626. No abstract available. PMID 12362012
- [Background] Rakvag TT, Klepstad P, Baar C, Kvam TM, Dale O, Kaasa S, Krokan HE, Skorpen F. The Val158Met polymorphism of the human catechol-O-methyltransferase (COMT) gene may influence morphine requirements in cancer pain patients. Pain. 2005 Jul;116(1-2):73-8. doi: 10.1016/j.pain.2005.03.032. PMID 15927391
- [Background] Nackley AG, Tan KS, Fecho K, Flood P, Diatchenko L, Maixner W. Catechol-O-methyltransferase inhibition increases pain sensitivity through activation of both beta2- and beta3-adrenergic receptors. Pain. 2007 Apr;128(3):199-208. doi: 10.1016/j.pain.2006.09.022. Epub 2006 Nov 7. PMID 17084978
- [Background] Diatchenko L, Nackley AG, Slade GD, Bhalang K, Belfer I, Max MB, Goldman D, Maixner W. Catechol-O-methyltransferase gene polymorphisms are associated with multiple pain-evoking stimuli. Pain. 2006 Dec 5;125(3):216-224. doi: 10.1016/j.pain.2006.05.024. Epub 2006 Jul 11. PMID 16837133
- [Background] Chou WY, Yang LC, Lu HF, Ko JY, Wang CH, Lin SH, Lee TH, Concejero A, Hsu CJ. Association of mu-opioid receptor gene polymorphism (A118G) with variations in morphine consumption for analgesia after total knee arthroplasty. Acta Anaesthesiol Scand. 2006 Aug;50(7):787-92. doi: 10.1111/j.1399-6576.2006.01058.x. PMID 16879459
- [Background] Klepstad P, Rakvag TT, Kaasa S, Holthe M, Dale O, Borchgrevink PC, Baar C, Vikan T, Krokan HE, Skorpen F. The 118 A > G polymorphism in the human mu-opioid receptor gene may increase morphine requirements in patients with pain caused by malignant disease. Acta Anaesthesiol Scand. 2004 Nov;48(10):1232-9. doi: 10.1111/j.1399-6576.2004.00517.x. PMID 15504181
- [Background] Reyes-Gibby CC, Shete S, Rakvag T, Bhat SV, Skorpen F, Bruera E, Kaasa S, Klepstad P. Exploring joint effects of genes and the clinical efficacy of morphine for cancer pain: OPRM1 and COMT gene. Pain. 2007 Jul;130(1-2):25-30. doi: 10.1016/j.pain.2006.10.023. Epub 2006 Dec 6. PMID 17156920
- [Background] Coulbault L, Beaussier M, Verstuyft C, Weickmans H, Dubert L, Tregouet D, Descot C, Parc Y, Lienhart A, Jaillon P, Becquemont L. Environmental and genetic factors associated with morphine response in the postoperative period. Clin Pharmacol Ther. 2006 Apr;79(4):316-24. doi: 10.1016/j.clpt.2006.01.007. PMID 16580900
- [Background] Coller JK, Barratt DT, Dahlen K, Loennechen MH, Somogyi AA. ABCB1 genetic variability and methadone dosage requirements in opioid-dependent individuals. Clin Pharmacol Ther. 2006 Dec;80(6):682-90. doi: 10.1016/j.clpt.2006.09.011. PMID 17178268
- [Background] Ikeda K, Ide S, Han W, Hayashida M, Uhl GR, Sora I. How individual sensitivity to opiates can be predicted by gene analyses. Trends Pharmacol Sci. 2005 Jun;26(6):311-7. doi: 10.1016/j.tips.2005.04.001. PMID 15925706
- [Background] Ameyaw MM, Regateiro F, Li T, Liu X, Tariq M, Mobarek A, Thornton N, Folayan GO, Githang'a J, Indalo A, Ofori-Adjei D, Price-Evans DA, McLeod HL. MDR1 pharmacogenetics: frequency of the C3435T mutation in exon 26 is significantly influenced by ethnicity. Pharmacogenetics. 2001 Apr;11(3):217-21. doi: 10.1097/00008571-200104000-00005. PMID 11337937
- [Background] Kim RB, Leake BF, Choo EF, Dresser GK, Kubba SV, Schwarz UI, Taylor A, Xie HG, McKinsey J, Zhou S, Lan LB, Schuetz JD, Schuetz EG, Wilkinson GR. Identification of functionally variant MDR1 alleles among European Americans and African Americans. Clin Pharmacol Ther. 2001 Aug;70(2):189-99. doi: 10.1067/mcp.2001.117412. PMID 11503014
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] von Baeyer CL, Spagrud LJ, McCormick JC, Choo E, Neville K, Connelly MA. Three new datasets supporting use of the Numerical Rating Scale (NRS-11) for children's self-reports of pain intensity. Pain. 2009 Jun;143(3):223-227. doi: 10.1016/j.pain.2009.03.002. Epub 2009 Apr 8. PMID 19359097
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Ramsay MA. Anesthesia and pain management at Baylor University Medical Center. Proc (Bayl Univ Med Cent). 2000 Apr;13(2):151-65. doi: 10.1080/08998280.2000.11927660. No abstract available. PMID 16389370
- [Background] Musani SK, Shriner D, Liu N, Feng R, Coffey CS, Yi N, Tiwari HK, Allison DB. Detection of gene x gene interactions in genome-wide association studies of human population data. Hum Hered. 2007;63(2):67-84. doi: 10.1159/000099179. Epub 2007 Feb 2. PMID 17283436
- [Background] Kelly PJ, Stallard N, Whittaker JC. Statistical design and analysis of pharmacogenetic trials. Stat Med. 2005 May 30;24(10):1495-508. doi: 10.1002/sim.2052. PMID 15706636
- [Background] Moore JH, Williams SM. New strategies for identifying gene-gene interactions in hypertension. Ann Med. 2002;34(2):88-95. doi: 10.1080/07853890252953473. PMID 12108579
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Park MY, Hastie T. Penalized logistic regression for detecting gene interactions. Biostatistics. 2008 Jan;9(1):30-50. doi: 10.1093/biostatistics/kxm010. Epub 2007 Apr 11. PMID 17429103
- [Background] Moons KG, Donders AR, Steyerberg EW, Harrell FE. Penalized maximum likelihood estimation to directly adjust diagnostic and prognostic prediction models for overoptimism: a clinical example. J Clin Epidemiol. 2004 Dec;57(12):1262-70. doi: 10.1016/j.jclinepi.2004.01.020. PMID 15617952
- [Background] Huth MM. Pediatric day surgery outcomes management: the role of preoperative anxiety and a home pain management protocol. J Child Fam Nurs. 1999 Jul-Aug;2(4):273-5. No abstract available. PMID 10646358